CLINICAL TRIAL: NCT04280016
Title: The Effect of Exercise on Wound Healing in People With Diabetes Undergoing Off-loading Treatment
Brief Title: The Effect of Exercise on Wound Healing While Off-loading
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mercer University (Other)
Responsible Party: Principal Investigator, Deborah M. Wendland, Ph.D., Associate Professor, Mercer University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H1908192
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes; off-loading; exercise
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A pilot study using retrospective chart review and non-randomized controlled trial methodology (single group).
Masking Description: The outcome assessor will be unaware of how much the participant participated in the exercise program. Exercise will occur away from the treatment area so that the care provider will be unaware of whether or not a patient is participating in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Added to Off-loading (Experimental): Participants in this arm will participate in exercise at the healthcare facility one time a week (away from where wound care is provided) and be instructed in a home exercise program that they will be encouraged to perform at least three days per week with no more than two days between sessions. Wound care will continue at the facility as is standard, utilizing off-loading.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Participants will participate in an exercise session with non-weight-bearing exercise that the participant is able to perform with off-loading (e.g. total contact cast) intact. They will also be instructed in a home exercise program so that exercise can be performed three days per week with no more than two days between sessions. These participants will also receive standard wound care with off-loading.

SUMMARY:
This study seeks to establish the effect of adding exercise to off-loading interventions on the healing time for people with diabetes mellitus and a foot ulcer. Hypothesis: Consistent with the literature, results are expected to resemble the accelerated healing seen when older adults exercised in the presence of wounds.

DETAILED DESCRIPTION:
The purpose of this project is to establish the effect of the addition of exercise to an off-loading intervention on the healing time for people with diabetes mellitus and a foot ulcer.

While benefits of physical activity and exercise are clear, the benefit of exercise on wound healing in individuals with diabetes has not been elucidated. It is critical to better understand how prescribed exercise effects the healing speed in patients receiving wound care with appropriate off-loading. If exercise does decrease healing time, the benefit to the patient may include lower cost, decreased risk of infection, decreased burden on a caregiver, and improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Have diabetes
* Have an active plantar ulceration
* With or without peripheral neuropathy
* Able to safely exercise
* Receiving care for their plantar ulceration, including off-loading

Exclusion Criteria:

- Presence of an untreated infection, osteomyelitis, or gangrene

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-05-14 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Wound measurement size | Measurements of wound will be taken up to 12 weeks or until wound closure occurs, whichever is first.
  Charts will be reviewed for normal wound measurements as is part of standard care. Measurements are expected to be reported as surface area (cm^2) and/or volume (cm^3). Wound closure will be defined as epithelialization across the entire wound bed and would be expected to correlate to no surface area or volume of wound being reported.

SECONDARY OUTCOMES:
Summary of Diabetes Self-Care Activities Scale | Measurement will be taken at baseline and at end of study (at 12 weeks or at wound closure, whichever occurs first).
  Participation in exercise. Using two questions, this scale measures the number of days that an individual reports doing physical activity (question 1) or specific exercise (question 2). Scores on each question could range from 0 to 7 days. The higher the number, the more days the individual participates in the activity or exercise.
Body Mass Index | Measurement will be taken at baseline and at end of study (at 12 weeks or at wound closure, whichever occurs first).
  Height and weight measurements will be combined and reported as BMI and measured in kg/m^2.
Physical activity data using an activity monitor (e.g. StepWatch). | Measured at baseline for one week.
  A week-long measurement of strides will be taken at the begin of the study.
Vibration sense | Measurement will be taken at baseline and at end of study (at 12 weeks or at wound closure, whichever occurs first).
  Vibration sense will be measured using a Bio-Thesiometer to assess for degree of peripheral neuropathy. A higher score would indicate decreased sensory perception of vibration.
Waist circumference | Measurement will be taken at baseline and at end of study (at 12 weeks or at wound closure, whichever occurs first).
  Waist circumference will be taken in cm as a marker of body composition.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah M. Wendland, Principal Investigator — Mercer University
Locations (1):
- Piedmont Healthcare, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified closure rate data will be made available through a repository upon conclusion of the study and its dissemination.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available following the study conclusion and its dissemination (6 months after publication).
Access Criteria: The information will be shared with researchers for meta-analyses through the data repository.